CLINICAL TRIAL: NCT01810640
Title: Pre-recovery Percutaneous Biopsy of Livers in Neurological Death Organ Donors - A Pilot Study
Brief Title: Pre-recovery Bedside Liver Biopsy in Brain Death Organ Donors
Acronym: PPB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Complications encountered with biopsy in first 6 patients
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Baburao Koneru, MD, Professor of Surgery, Division Chief Liver Transplantation, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012002002
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Brain Death; Liver Disease
Keywords: Liver biopsy; organ donation; donor management
MeSH Terms: conditions — Brain Death; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): In this group a liver biopsy will not be performed. All management would be as per standard of practice
- Percutaneous liver biopsy (Active Comparator): In this group a percutaneous biopsy of the liver will be performed prior to organ recovery
  Interventions: Procedure: Percutaneous Liver Biopsy

INTERVENTIONS:
Procedure: Percutaneous Liver Biopsy — Using a 16 gauge Jamshidi biopsy needle, without image guidance, 3 passes will be completed to obtain core liver biopsies. Biopsies will be placed on wet saline and processed via frozen sample in OCT compound in 5 micron slices and stained with hematoxylin and eosin for microscopic evaluation. Slides will then be digitalized and shared on Donor.net.
  Other Names: Bedside Liver Biopsy
  Arms: Percutaneous liver biopsy

SUMMARY:
This study's objective is to obtain preliminary data to test the hypotheses that percutaneous liver biopsy in brain death donors is safe and provides reliable histological information. Furthermore, that information when disseminated fully and widely many hours before organ recovery would not only decrease economic costs of wasteful recovery of livers that are not ultimately transplanted but also increase transplantation and decrease cold ischemia times of recovered livers.

ELIGIBILITY:
Inclusion Criteria:

* Neurological death donors in whom brain death determination is imminent
* First person or next of kin consent for research becomes available
* High risk donor, as defined by the following criteria i) Known liver disease ii) Hepatitis BsAg, BcAb, B DNA, Hepatitis C Ab or Hepatitis C RNA positivity iii) Age >= 50 iv) Any of the following risk factors for fatty liver disease a) BMI >= 30 b) History of Type 2 Diabetes Mellitus c) Ultrasound, Computerized Tomography or other imaging modalities suggesting steatosis v) Any of the following risk factors for chronic liver disease

  1. Greater than 2 drinks of alcohol daily currently or in their history
  2. Current IV drug use
  3. Ultrasound, Computerized Tomography or other imaging modalities suggesting cirrhosis

Exclusion Criteria:

* Donation after cardiac death donors
* Live organ donors
* No first person consent and next of kin decline research consent
* Donors in whom it has been established the liver will not be shared
* Donors in whom percutaneous liver biopsy has been performed within the past month for any indication and the biopsy results are available and considered reliable.
* Donor with a contraindication to liver biopsy, including INR > 2, PTT > 75, Platelets < 70,000, history of coagulopathy, current or recent use (within 7 days) of antiplatelet agent such as aspirin or Plavix, and hemodynamic instability defined as a MAP less than 65mmHg.
* Inability to position donor appropriately for performance of PPB
* Unavailability of pathology staff to analyze specimen in a timely manner

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety | 6 hours
  Safety of bedside liver biopsy will be measured as the presence or absence of a composite outcome of: change in hemoglobin (gm/dL) from baseline of greater than 2, occurence of pneumothorax on right side observed on chest X-ray immediately after biopsy, and/or donor instability leading to expedited organ recover, and/or loss of donor organs attributed to the biopsy
Reliability | 24hrs
  Agreement of the findings of the bedside biopsy with reference to an intraoperative biopsy in histological characteristics of steatosis, inflammation, and fibrosis
Feasibility | 24hrs
  The proportion of donors in the biopsy group in whom PPB information becomes available prior to commencement of organ recovery

SECONDARY OUTCOMES:
Feasibility | 24hrs
  Time between performance of biopsy and availability of results to the sharing network

CONTACTS AND LOCATIONS:
Overall Officials: Babuaro Koneru, MD, Principal Investigator — UMDNJ - New Jersey Medical School
Locations (2):
- United States (2):
  - New Jersey Organ and Sharing Network, New Providence, New Jersey
  - University Hospital, Newark, New Jersey